CLINICAL TRIAL: NCT06741176
Title: The Effect of the Message Left by Mothers Whose Babies Are in the Neonatal Intensive Care Unit to Their Babies on Mother-Baby Attachment and Hope Level: Randomized Controlled Study
Brief Title: The Effect of the Message Left by Mothers Whose Babies Are in the Neonatal Intensive Care Unit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semra Kose (Other)
Responsible Party: Sponsor-Investigator, Semra Kose, Assistant Professor (PhD, RN), Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NEU2024breastmilk
Record Dates: First submitted 2024-12-16; First posted 2024-12-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Breast Milk; Premature
Keywords: Premature; breast milk; Mother; attachment; Hope
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled trial in experimental design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Triple (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Breast Milk
  Interventions: Behavioral: Experimental
- Control (Active Comparator): Control
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Experimental — The research data will be collected with mothers whose babies are in the NICU. Information about the research will be given to mothers who come to leave milk for their babies and the research will be conducted with those who agree to participate. All surveys will be pre-tested on the mothers without randomization and the group they are in will be determined by randomization. The mothers in the experimental group will be asked to write messages to their babies on the milk bags they bring in the mornings for 3 days. They will be asked to write on the paper attached to the milk bag what they want to tell their baby that the investigators will read the message to them and to return it every morning. The post-test of all surveys will be conducted at the end of the 3rd day.
  Arms: Experimental
Behavioral: Control — The research data will be collected with mothers whose babies are in the NICU. Information about the research will be given to mothers who come to leave milk for their babies and the research will be conducted with those who agree to participate. All surveys will be pre-tested on the mothers without randomization and the group they are in will be determined by randomization. The post-tests will be conducted 3 days after the pre-test without any messages being requested from the mothers in the control group.
  Arms: Control

SUMMARY:
Newborn babies may need to stay in neonatal intensive care units (NICU) immediately after birth for many reasons such as premature birth, low birth weight, respiratory distress, infection, jaundice. Depending on the cause and level of the newborn's illness, the length of stay may be extended, lasting weeks or even months. This situation negatively affects mother-infant bonding, causing mothers to be unable to establish healthy communication with their babies. For mothers in particular, leaving their babies in the NICU makes them feel inadequate and hopeless.

Attachment is the emotional bond that a baby establishes with its mother or the person who cares for it. This bond established between the mother and the baby affects the emotional, social, cognitive and moral development of the individual throughout their life. It is known that secure attachment contributes to the physical and mental development of babies, while insecure attachment is associated with various mental illnesses. For these reasons, it is important to initiate secure attachment between the mother and the baby during the neonatal period.

The aim of this planned study is to examine the effect of the messages left by mothers whose babies are in the NICU on mother-infant bonding and the mothers' level of hope. Mothers leaving messages for their babies provides a context in which they can express themselves to their babies and may positively affect mother-infant bonding and the mother's level of hope in the NICU.

DETAILED DESCRIPTION:
Babies in the first four weeks (0-28 days) after birth are called newborns. The newborn period is a high-risk period for babies, and during this period, newborns need optimal care to survive. In 2018, 2.5 million newborns lost their lives due to preventable causes. NICUs are intensive care units equipped with high technology to meet all the needs of newborns; consisting of neonatologists, neonatologists and neonatal intensive care nurses. There may be many reasons for a baby to be admitted to the NICU. Some of these are; premature birth, low birth weight, respiratory distress, infection, jaundice, malnutrition, perinatal hypoxia, congenital heart disease, metabolic disorders and other congenital anomalies. While the baby's stay in the intensive care unit is necessary for its vital functions, this process also negatively affects the mother-baby bonding process. The mother breastfeeding her baby, ensuring early skin-to-skin contact, staying in the same room, the process of getting used to the role of motherhood, the social support the mother receives after birth are some of the factors that affect mother-baby bonding. The hospitalization of a baby disrupts the mother-baby relationship and can harm the mental health of parents and the development of babies. Parents face problems such as hopelessness, stress, psychological distress, loss of parental role and disruption of mother-baby bonding. The hospitalization of a baby in the NICU creates a traumatic effect on the family and disrupts bonding. Therefore, it is important to effectively initiate and develop mother-baby bonding for the health and future of the mother and baby. Hope is a dynamic force that empowers the individual to adapt to the future, enables them to be interested in their current life and the future and find meaning in it, supports well-being and helps maintain relationships with others. The lack of knowledge about the diagnosis and treatment procedures of babies admitted to neonatal units, the uncertainty of the prognosis, the reactions of the baby and most importantly, the lack of sufficient explanations from healthcare professionals can be shown as factors that lead to hopelessness in mothers. Other factors that increase hopelessness are the mother's inability to decide when to visit her baby, when to see the doctor and when to get information from healthcare professionals. The neonatal nurses who accept the baby can play an active role in the hope of the mother whose baby is hospitalized for her baby to grow and develop healthily. Creating a comfortable environment during the admission where the mother will perceive herself as a part of the unit rather than a visitor, welcoming the baby and the family, the nurse who will care for the baby introducing herself to the family, showing the place where the baby will stay and introducing the unit and providing information about this can reduce the anxiety and fear of the parents and the hopelessness of the mother who cannot hold her baby in her arms and breastfeed. On the other hand, mothers being with their babies and participating in their care at the earliest possible stage in this process can contribute to the bonding process, the growth and development of the baby, and the reduction of parents' hopelessness regarding their babies and the development of their problem-solving skills regarding baby care. Although there are studies in the literature on the hopelessness levels of mothers receiving care in the NICU and on mother-infant attachment in the NICU, no randomized controlled study has been found that included mothers leaving messages for their babies. Therefore, the aim of the planned study was to examine the effects of the messages left by mothers whose babies are in the NICU on mother-infant attachment and the mothers' level of hope.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the care of the baby,
* Reading and understanding Turkish,

Exclusion Criteria:

- No psychological problems in the mother

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic Information Form | It will be applied to mothers who are breastfeeding for the first time by the researcher (approximately 5 minutes)
  The form, which was developed by the researcher by scanning the literature, has a total of 16 questions. It includes questions such as the mother's age, occupation, education level, baby's gender, weight, and week of birth.
Mother-Infant Bonding Scale | Mothers who are breastfeeding for the first time will fill it out themselves on the first day (pre-test) and the 3rd day (post-test). (approximately 10 minutes)
  The eight-item scale filled out by the mother consists of eight items that include the emotional states the mother feels towards her baby after birth. The scale items consist of a four-point Likert-type rating, from "(0) very much" to "(3) never". Five items indicating negative emotions are scored in reverse (3-0). A high score indicates that the mother and baby have a bonding problem. The internal consistency coefficient of the scale was reported as 0.66 in the validity and reliability study.
State Hope Scale | Mothers who are breastfeeding for the first time will fill it out themselves on the first day (pre-test) and the 3rd day (post-test). (approximately 10 minutes)
  The Turkish validity and reliability study of the State Hope Scale developed by Snyder et al. (1996) was conducted by Bekmezci et al. (2021). The statements in the Hope Scale were measured with an eight-point Likert (1=Absolutely false, 8=Absolutely true). The State Hope Scale consists of 2 dimensions: active thought and the ability to think of alternative ways to reach the goal. Questions 1, 3 and 5 in the scale measure the ability to think of alternative ways to reach the goal; questions 2, 4 and 6 measure the active thought dimension. High scores from the dimensions indicate high hope.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No